CLINICAL TRIAL: NCT06541223
Title: Effect of a Multimedia-assisted Informed Consent Procedure on the Information Gain, Satisfaction and Anxiety of Patients Undergoing Mastectomy and Implant-based Reconstruction
Brief Title: Multimedia-assisted Informed Consent Procedure for Patients Undergoing Mastectomy and Implant-based Reconstruction
Status: Completed | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1999
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; High-risk healthy patients; Implant-based reconstruction; Multimedia-assisted informed consent procedure
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard Informed Consent Procedure: Face-to-face informed consent procedure supported by an informational brochure approved by the hospital committee
  Interventions: Other: Standard informed consent procedure
- Multimedia Assisted Informed Consent Procedure: Face-to-face informed consent procedure supported by an informational brochure approved by the hospital committee, followed by a multimedia presentation on implant-based reconstruction
  Interventions: Other: Standard informed consent procedure; Other: Multimedia video

INTERVENTIONS:
Other: Standard informed consent procedure — Face-to-face informed consent procedure supported by informational brochure
Other: Multimedia video — Multimedia presentation on implant-based reconstruction
  Groups: Multimedia Assisted Informed Consent Procedure

SUMMARY:
Breast reconstruction is a women's right with positive psychological effects and it is an integral part of breast cancer treatment and care. A preoperative counselling is mandatory, providing information about oncologic surgery, the type of reconstruction and the expected results. This study plans to compare conventional informed consent process supported by informational brochures with a multimedia video-assisted procedure supported by the same informational brochures in breast cancer patients undergoing immediate implant-based reconstruction. The two processes will be compared in terms of information retention, patient satisfaction of the informed consent process and anxiety levels before surgery.

DETAILED DESCRIPTION:
Implant-based reconstruction is the most frequent procedure after mastectomy, able to preserve body integrity and femininity. Breast reconstruction is a women's right with positive psychological effects. It is an integral part of breast cancer treatment and care, and in the vast majority of cases it is performed in the immediate setting. Breast reconstruction is personalized and tailored to each patient, taking in consideration patient anatomy and comorbidities, cancer staging and oncologic rules and even patient desires. Patient expectations are very high and women are seeking for outstanding cosmetic results especially in case of prophylactic surgery, therefore preoperative counselling is mandatory, providing information about oncologic surgery, the type of reconstruction and the expected results. A detailed informed consent procedure must include explanations of the surgical procedure, including its benefits, alternatives and risks, information about the implants (temporary or definitive ones) and postoperative scenarios. The face-to-face discussion is supported by information brochures that include all this information. Unfortunately, the readability of these documents is often not high and the rate of information retention might be low. Recently, it has been observed that the amount of information retained by patients appears to improve using a multi-media video-assisted informed consent procedure. Aim of this study is to evaluate if a multimedia-assisted video tutorial before implant-based reconstruction could increase the information retained by patients, their satisfaction about the informed consent process and influence their anxiety levels before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing mastectomy for breast cancer
* High-risk healthy patients undergoing risk reducing mastectomies
* Unilateral and/or bilateral mastectomies
* If unilateral mastectomy, both patients requiring or not contralateral mammaplasty of the healthy breast

Exclusion Criteria:

* Patients undergoing mastectomy and autologous reconstruction
* Patients who previously underwent unilateral mastectomy and implant reconstruction, requiring contralateral mastectomy
* Patients not available for e-correspondence

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing mastectomy and implant-based reconstruction (both with definitive implants and temporary prostheses or expanders)
Sampling Method: Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of current state of anxiety | 2 weeks
  Collection of Spielberger State/Trait Anxiety Inventory (STAI) Y1 questionnaire (minimum value: 1, maximum value: 4 - higher scores mean greater anxiety)
Evaluation of anxiety proneness | 2 weeks
  Collection of Spielberger State/Trait Anxiety Inventory (STAI) Y2 questionnaire (minimum value: 1, maximum value: 4 - higher scores mean greater anxiety)
Evaluation of uncertainty and perceptions of effective decision-making | 2 weeks
  Collection of Decisional Conflict Scale (DCS) questionnaire (minimum value: 1, maximum value: 5 - higher scores mean higher decisional conflict)
Evaluation of patients' understanding of plastic reconstruction procedures and surgical complications | 2 weeks
  Collection of Reconstructive Breast Surgery Comprehension Questionnaire (minimum value: 1, maximum value: 4 - higher scores mean better understanding)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca De Lorenzi, MD, Principal Investigator — European Istitute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy